CLINICAL TRIAL: NCT00504621
Title: The Influence of Personality on Quality of Life, Fatigue, Prognosis, and Health Care Consumption in Pulmonary Fibrosis and Sarcoidosis
Brief Title: The Influence of Personality on Pulmonary Fibrosis and Sarcoidosis
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Tilburg University (Other)
Responsible Party: Sponsor
Other Study IDs: MEC 07-4-015
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Sarcoidosis; Pulmonary Fibrosis
Keywords: personality; fatigue; quality of life; health care consumption
MeSH Terms: conditions — Sarcoidosis; Pulmonary Fibrosis; Fatigue

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- sarcoidosis: Sarcoidosis known by the ild care team of the outpatient clinic of the department of Respiratory Medicine of the University Hospital Maastricht as well as new patients attending the out-patient clinic from August 2007 to January 2009
- pulmonary fibrosis: Idiopathic pulmonary fibrosis (IPF) patients known by the ild care team of the outpatient clinic of the department of Respiratory Medicine of the University Hospital Maastricht as well as new patients attending the out-patient clinic from August 2007 to January 2009

SUMMARY:
A number of studies have shown that the quality of life of two common interstitial lung diseases (ild), sarcoidosis and pulmonary fibrosis patients, is impaired and that fatigue is a substantial problem for those patients. Furthermore, breathlessness is an additional major problem in pulmonary fibrosis. In the field of cardiovascular disease and breast cancer, personality factors have shown to play a role in patient's morbidity, mortality, quality of life, fatigue, depressive symptoms, and one study showed a predictive role of personality factors in health care consumption. No studies examining personality factors have been performed in sarcoidosis or pulmonary fibrosis. Therefore, the aim of the present study is to examine the role of personality factors as predictors of fatigue, quality of life, prognosis, and health care consumption in sarcoidosis and pulmonary fibrosis. In this study a number of possible moderators, such as social support, will also be examined, aiming to get a full picture of the relationship between the various factors examined. Known and new sarcoidosis and pulmonary fibrosis patients (inclusion period 1 year) of ild care team of the outpatient clinic of the department of Respiratory Medicine of the University Hospital Maastricht will be asked to participate through completing questionnaires at baseline and every six months for 18 months, and allowing the researchers access to their medical records for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to be diagnosed with sarcoidosis based on consistent clinical features and BAL fluid analysis results, according to the WASOG guidelines.
* The diagnosis IPF will be made based on the ATS guidelines

Exclusion Criteria:

* Poor expression in the Dutch language
* Relevant co morbidity such as a malignancy, dementia, and a history of psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sarcoidosis patients diagnosed according to WASOG guidelines and IPF patients diagnosed according ATS guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The role of personality factors as predictors in sarcoidosis and pulmonary fibrosis. | 18 months
  The role of personality factors as predictors of fatigue, quality of life, prognosis, and health care consumption in sarcoidosis and pulmonary fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Drent, Md, PhD, Study Chair — Maastricht University; Jolanda de Vries, PhD, Study Chair — Tilburg University; Marjon Elfferich, MSc, Principal Investigator — Gelderse Vallei Ziekenhuis Ede

REFERENCES:
- [Result] Elfferich MD, De Vries J, Drent M. Type D or 'distressed' personality in sarcoidosis and idiopathic pulmonary fibrosis. Sarcoidosis Vasc Diffuse Lung Dis. 2011 Jul;28(1):65-71. PMID 21796893